CLINICAL TRIAL: NCT03833024
Title: The MUFFIN-PTS Trial: Micronized Purified Flavonoid Fraction for the Treatment of Post-Thrombotic Syndrome
Brief Title: The MUFFIN-PTS Trial
Acronym: MUFFIN-PTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Susan Kahn, Professor of Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 332593-S1
Record Dates: First submitted 2019-01-30; First posted 2019-02-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Post-Thrombotic Syndrome
Keywords: deep vein thrombosis; chronic venous insufficiency; venoactive drug; Micronized Purified Flavonoid Fraction; DVT; post thrombotic syndrome
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo-controlled trial with oral placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venixxa (Active Comparator): Micronized Purified Flavonoid Fraction (MPFF) for 6 months MPFF 500 mg, BID (morning and evening) for 6 months
  Interventions: Drug: Micronized Purified Flavonoid Fraction
- Placebo (Placebo Comparator): Placebo for 6 months
  1 Tablet, BID (morning and evening) for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Micronized Purified Flavonoid Fraction — After randomization (1:1 with stratification by centre) patients will receive 1000 mg of oral MPFF (Venixxa, one 500mg tablet BID) for 6 months, in addition to their usual PTS and DVT treatment
  Other Names: Venixxa group
  Arms: Venixxa
Drug: Placebo — After randomization (1:1 with stratification by centre) patients will receive an oral placebo (one tablet BID) for 6 months, in addition to their usual PTS and DVT treatment
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
In this randomized controlled trial (RCT), the investigators will determine whether a 6-month course of oral Micronized Purified Flavonoid Fraction (MPFF 1000 mg daily), compared with placebo, improves the symptoms and signs of the post-thrombotic syndrome (PTS) and quality of life (QOL) at 6 months follow-up.

DETAILED DESCRIPTION:
The post thrombotic syndrome (PTS) is a form of secondary chronic venous insufficiency (CVI) that develops after a deep vein thrombosis (DVT). It affects up to 50% of patients after a proximal DVT (i.e. DVT involving popliteal vein or more proximal veins), and 5-10% of patients develop severe PTS. PTS is a chronic condition that reduces quality of life (QOL) and for which no curative treatment is available. Cornerstones of PTS treatment include the use of elastic compression stockings (ECS) to reduce leg symptoms and prevent PTS progression. However, ECS are incompletely effective, burdensome and costly to patients. Micronized Purified Flavonoid Fraction (MPFF, Venixxa), a venoactive drug, has been reported to be effective in reducing venous symptoms and signs and improving QOL in patients with CVI and has the potential to be effective for the treatment of PTS. Further, use of Venixxa is safe, with only few very mild and reversible reported side effects. However, studies of MPFF in patients with CVI have been of low to moderate quality, and there has been little use of this drug in North America. In addition, the effectiveness of MPFF has never been specifically evaluated in patients with PTS. Given that the pathophysiological mechanism of PTS is complex and unique (combination of obstructive and reflux mechanisms as well as inflammation), it is uncertain if MPFF is effective in patients with PTS, even if it may be effective for CVI more generally.

The MUFFIN-PTS study will be a multicentre (8-10 centres), randomized, placebo-controlled trial. Patients will be randomized (1:1 with stratification by centre) to receive 1000 mg of oral MPFF (Venixxa, one 500mg tablet BID) or an identically appearing placebo (one tablet BID) for 6 months, in addition to their usual PTS and DVT treatment (i.e. ECS and/or anticoagulation, at their treating physician's discretion). Its objectives are to evaluate the effectiveness and safety of MPFF (Venixxa) compared to placebo for the treatment of PTS.

86 patients with lower limb PTS will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Villalta score ≥5 with at least two of the following four PTS manifestations (daily heaviness, cramps, pain, and objective edema) in the leg ipsilateral to a previous objectively diagnosed DVT, or DVT of unknown date but with presence of residual proximal or distal venous obstruction on ultrasound. Females of childbearing age must use medically approved method of birth control and must have negative pregnancy test results at the time of randomization.

Exclusion Criteria:

* Recent acute ipsilateral DVT (<3 months)
* Active ipsilateral venous ulcer
* Acute or chronic altered mental status
* Any venoactive drug intake within 3 months of the start of the study
* Allergy or hypersensitivity to MPFF/Venixxa
* Age<18 years
* Pregnant or breastfeeding women
* Life expectancy <1 year
* Refuse or unwilling to provide consent
* Unable to speak English or French
* Alcohol/drug abuse
* Hospitalized patients
* End-stage kidney disease (dialysis, creatinine clearance < 10ml/min)
* Liver cirrhosis Child-Pugh class C.
* Currently enrolled in other clinical trials, other than trials of prevention or treatment of venous thromboembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in PTS | 6 months
  Improvement will be defined as a decrease of at least 30% in the Villalta score or a Villalta score <5 in the PTS-affected leg.

SECONDARY OUTCOMES:
Severity of PTS | baseline, 3, 6 and 9 months
  Villalta score category (mild, moderate, severe)
Change in PTS | 3 and 9 months
  Improvement will be defined as a decrease of at least 30% in the Villalta score or a Villalta score <5 in the PTS-affected leg.
Venous specific Quality of life | 3, 6 and 9 months
  Venous-disease specific (VEINES-QOL) score
General Quality of life | 3, 6 and 9 months
  Generic QOL (EQ-5D-5L) score. The EQ-5D-5L consists of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.
Serious Adverse Events (SAE) | 9 months
  Includes drug-related SAE, DVT, Pulmonary Embolism (PE), death
Patient compliance with treatment | 3 and 6 months
  Judged satisfactory if at least 80% of the study drug was reportedly taken
Patients' overall satisfaction with treatment | 3 and 6 months
  Assessed with a 5-point Likert visual analog scale questionnaire (1 indicate patient is very satisfied with treatment and 5 that he is very unsatisfied)
Villalta score | 3, 6, 9 months
  Villalta score assessed as a continuous variable (greater score indicates more severe disease, score range 0 to 33)
Pain as a symptom of PTS | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Cramps | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Heaviness | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Paresthesia | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Pruritus | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Pre-tibial edema | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Hyperpigmentation | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Redness | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Skin induration | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Venous ectasia | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent to 3 severe)
Venous Ulcer | 3, 6, 9 months
  Analyzed as individual component of Villalta score (0 absent or 1 present)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Kahn, MD, MSc, Principal Investigator — Jewish General Hospital (Montreal, Quebec, Canada); Jean-Philippe Galanaud, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
Locations (7):
- Canada (7):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Open access to individual patient data is not planned, but all requests for the trial's data will be considered on an individual basis by the trial steering committee

REFERENCES:
- [Background] Kahn SR, Pengo V. Special issue: Late consequences of venous thromboembolism. Thromb Res. 2018 Apr;164:99. doi: 10.1016/j.thromres.2018.02.005. Epub 2018 Feb 13. No abstract available. PMID 29459016
- [Background] Rabinovich A, Kahn SR. How I treat the postthrombotic syndrome. Blood. 2018 May 17;131(20):2215-2222. doi: 10.1182/blood-2018-01-785956. Epub 2018 Mar 15. PMID 29545327
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Background] Galanaud JP, Monreal M, Kahn SR. Epidemiology of the post-thrombotic syndrome. Thromb Res. 2018 Apr;164:100-109. doi: 10.1016/j.thromres.2017.07.026. Epub 2017 Jul 24. PMID 28844444
- [Background] Cohen JM, Akl EA, Kahn SR. Pharmacologic and compression therapies for postthrombotic syndrome: a systematic review of randomized controlled trials. Chest. 2012 Feb;141(2):308-320. doi: 10.1378/chest.11-1175. PMID 22315114
- [Background] Martinez-Zapata MJ, Vernooij RW, Uriona Tuma SM, Stein AT, Moreno RM, Vargas E, Capella D, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2016 Apr 6;4(4):CD003229. doi: 10.1002/14651858.CD003229.pub3. PMID 27048768
- [Background] Bush R, Comerota A, Meissner M, Raffetto JD, Hahn SR, Freeman K. Recommendations for the medical management of chronic venous disease: The role of Micronized Purified Flavanoid Fraction (MPFF). Phlebology. 2017 Apr;32(1_suppl):3-19. doi: 10.1177/0268355517692221. PMID 28211296
- [Background] Rabe E, Agus GB, Roztocil K. Analysis of the effects of micronized purified flavonoid fraction versus placebo on symptoms and quality of life in patients suffering from chronic venous disease: from a prospective randomized trial. Int Angiol. 2015 Oct;34(5):428-36. Epub 2015 May 14. PMID 25972136
- [Derived] Galanaud JP, Abdulrehman J, Lazo-Langner A, Le Gal G, Shivakumar S, Schulman S, Kahn S. MUFFIN-PTS trial, Micronized Purified Flavonoid Fraction for the Treatment of Post-Thrombotic Syndrome: protocol of a randomised controlled trial. BMJ Open. 2021 Sep 13;11(9):e049557. doi: 10.1136/bmjopen-2021-049557. PMID 34518263